CLINICAL TRIAL: NCT07209657
Title: A Parallel Mixed Methods Investigation of a Music Interventions in Paediatric Disorders of Consciousness (DoC)
Brief Title: Describing the Effect of Familiar Song on Arousal and Awareness for Children With Disorders of Consciousness (DoC)
Acronym: SongDoC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 113687
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Disorder of Consciousness; Acquired Brain Injury
Keywords: music therapy; music; paediatric disorder of consciousness
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries

STUDY DESIGN:
Intervention Model Description: This study is a single site, parallel mixed method incorporating a within subject design (trial).
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the interventions (recorded music vs live music therapy), the interventionist, participant, and parent/legal guardian cannot be masked. However, the investigator conducting the pre-post consciousness assessment (SECONDS) will be masked. The Research Assistant (RA) completes the pre-measure before the interventionist enters the room and the post-measure after the interventionist leaves, ensuring no overlap. The interventionist always carries equipment for both conditions to maintain concealment. Behavioural ratings from the video-recorded sessions will be completed with sound removed so the RA is masked to condition. Parents/caregivers are instructed not to reveal allocation; any unblinding will be logged and reported.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live music therapy intervention (Experimental): Live music therapy sessions will be delivered by an experienced music therapist using familiar songs with guitar accompaniment. Musical elements may be adapted in real time in response to the child's behaviours to support engagement. Each session will last about 20 minutes, tailored to the child's reduced state of consciousness and to minimise overstimulation or fatigue.
  Interventions: Behavioral: Live Music Therapy
- Recorded music intervention (Experimental): Recorded music interventions will use commercially available recordings of the same familiar songs presented in the live sessions, with only the format differing. The same music therapist will remain present in the room and play the recordings through an iPad and portable speaker.
  Interventions: Behavioral: Recorded Music

INTERVENTIONS:
Behavioral: Live Music Therapy — The recorded music interventions will consist of the presentation of commercially available recordings of participant preferred music. The songs utilised in the recorded music interventions will be the same as those presented during the live music therapy interventions, and only the presentation format will be different. The same music therapist who facilitates the live music therapy interventions will be present in the participant's room during the presentation of the recorded music intervention and will present the recorded music via iPad and small portable speaker.
  Arms: Live music therapy intervention
Behavioral: Recorded Music — The recorded music interventions will consist of the presentation of commercially available recordings of participant preferred music. The songs utilised in the recorded music interventions will be the same as those presented during the live music therapy interventions, and only the presentation format will be different. The same music therapist who facilitates the live music therapy interventions will be present in the participant's room during the presentation of the recorded music intervention and will present the recorded music via iPad and small portable speaker.
  Arms: Recorded music intervention

SUMMARY:
The goal of this clinical trial is to compare the effect of live music therapy and recorded music on recovery of consciousness in children aged 1 to 18 years who have a disorder of consciousness (DoC) after a severe brain injury. Researchers also want to learn how children respond during music and noise, whether early responses to music are linked to recovery at 6 months, and how parents experience music therapy during their child's hospital stay at The Royal Children's Hospital (RCH) in Melbourne.

Participants will:

* Take part in a 10-day study period while in hospital. On 8 of the 10 days, they will receive either live or recorded familiar music in random order. Their level of consciousness will be measured before and after each session using a simple behavioural checklist. On the other 2 days, they will take part in video-recorded sessions to compare behavioural responses during live music, recorded music, and white noise. Videos will help capture small changes in movement, eye gaze, or facial expression.
* Have their level of consciousness checked again at 6 months after injury to see if early responses relate to later recovery.

Parents and caregivers will be invited to take part in an interview about their experiences and observations of music therapy with their child.

This study will help researchers understand whether live music therapy provides benefits beyond recorded music and will guide how music therapy is best used to support children and families during recovery from severe brain injury.

DETAILED DESCRIPTION:
A disorder of consciousness (DoC) is a common consequence of severe acquired brain injury (ABI) in children. Children may present in coma, unresponsive wakefulness, or a minimally conscious state, and the duration of DoC is strongly linked with long-term recovery. Early, well-designed interventions are important to support emergence to consciousness and improve outcomes.

Music is considered a particularly meaningful stimulus for children because it is familiar, engaging, and closely linked with memory, emotion, and development. Live music therapy may offer additional benefits because the therapist can adjust the music in real time to the child's responses, potentially extending arousal and engagement. Recorded music, however, can be delivered more widely by families or healthcare staff, and may be more scalable. Despite widespread clinical use, especially at The Royal Children's Hospital (RCH) Melbourne, the scientific evidence for music therapy with children in DoC remains limited, and most prior studies have focused on adults.

This parallel mixed-method study has been designed to build robust paediatric-specific evidence through four integrated components:

Within-subject randomised trial (Component 1):

Participants will complete a 10-day data collection period during hospital admission.

On 8 of these days, participants will receive either live music therapy or recorded familiar music, with the order randomised.

Consciousness will be measured before and after each session using a paediatric adaptation of the Simplified Evaluation of Consciousness Disorders (SECONDS).

The objective is to determine whether live therapist-facilitated interventions are more effective than recorded interventions in supporting consciousness recovery.

Multiple baseline case series (Component 2):

On 2 of the 10 days, participants will take part in video-recorded sessions comparing responses during live music, recorded music, and white noise.

Behavioural responses (such as gaze, facial expression, and movement) will be coded to capture subtle and immediate changes that may not last long enough to appear in pre-post measures.

This component provides a mechanistic understanding of how children respond during auditory stimulation.

Six-month follow-up assessment (Component 3):

At 6 months post-injury, participants' level of consciousness will be reassessed in person or via telehealth.

This assessment will test whether early responsiveness to music interventions or behavioural responses during sessions are linked with longer-term recovery.

Parent and caregiver interviews (Component 4):

Parents and caregivers will be invited to take part in semi-structured interviews about their observations and experiences of music therapy during their child's admission.

Data will be analysed thematically to ensure family perspectives are embedded in the design of future clinical interventions.

Expected outcomes:

This study will provide the first controlled paediatric data comparing live and recorded music therapy in DoC. It will show whether live interventions provide unique benefits, whether early responsiveness predicts recovery, and how families experience music therapy during a critical stage of hospitalisation. Results will have immediate clinical translation by guiding how music interventions are best delivered and resourced, potentially supporting faster emergence to consciousness, shorter hospital stays, and improved wellbeing for children and their families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a severe ABI, as indicated by at least one of the following:

  * Glasgow Coma Scale (GCS) 3-8 at admission to RCH
  * Mass pathology evident on neuroimaging
  * Expert opinion of treating consultant
* Diagnosis of a DoC, as indicated by at least one of the following:

  * Rancho Los Amigos Scale I, II, III or IV
  * Expert opinion of treating consultant
* Legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf. Interpreters will be employed as necessary.

Exclusion Criteria:

* ABI not compatible with life/child expected to die
* ABI resulting from suspected non-accidental causes, including assault/abuse
* Diagnosed premorbid or acquired severe hearing loss
* Inability or unwillingness of legally acceptable representative to give written informed consent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Pre-post intervention change in the 'Simplified Evaluation of Consciousness Disorders (SECONDs)' | Days 1-2; 4-5; 6-7; 9-10, and at 6 months post-injury
  The Simplified Evaluation of Consciousness Disorders (SECONDS) is an 8-item behavioural scale assessing responsiveness across the spectrum of disorders of consciousness (DoC). Items progress in complexity from arousal response (1) to functional communication (8). The SECONDS is adapted from the Coma Recovery Scale-Revised but is faster to administer, making it suitable in acute paediatric settings. It has strong validity and inter-rater reliability in diagnosing prolonged DoC. For this trial, child-friendly modifications are used (e.g., age-appropriate toys, picture books, and yes/no questions) to ensure suitability for children.

SECONDARY OUTCOMES:
Changes in the 'Music interventions in paediatric DoC observation record (MBR)' outcomes across live music, recorded music, and control noise condition | Days 3 and 8
  The Music Behavioural Response Checklist (MBR) records behavioural responses during music interventions in children with disorders of consciousness (DoC). It has two sections: (1) arousal, capturing 13 discrete movement categories, and (2) awareness, capturing 15 categories of more complex behaviours linked to minimally conscious states and emergence. The MBR was developed and validated at the Royal Children's Hospital, showing content validity and fair to substantial inter-rater reliability. It is completed from video recordings to ensure subtle and idiosyncratic behaviours are captured.

CONTACTS AND LOCATIONS:
Overall Officials: Janeen M Bower, PhD, Principal Investigator — University of Melbourne
Locations (1):
- The Royal Children's Hospital Melbourne, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Pending extended consent from the participant's legal guardian, de-identified Individual Participant Data (IPD) will be made available for long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start date: 60 months following results dissemination via publication End date: When the youngest study participant turns 25 years of age
Access Criteria: IPD may be accessed by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre

REFERENCES:
- [Background] Molteni E, Canas LDS, Briand MM, Estraneo A, Font CC, Formisano R, Fufaeva E, Gosseries O, Howarth RA, Lanteri P, Licandro GI, Magee WL, Veeramuthu V, Wilson P, Yamaki T, Slomine BS; as the Special Interest Group on DoC of the International Brain Injury Association (IBIA-DoC SIG). Scoping Review on the Diagnosis, Prognosis, and Treatment of Pediatric Disorders of Consciousness. Neurology. 2023 Aug 8;101(6):e581-e593. doi: 10.1212/WNL.0000000000207473. Epub 2023 Jun 12. PMID 37308301
- [Background] Aubinet C, Cassol H, Bodart O, Sanz LRD, Wannez S, Martial C, Thibaut A, Martens G, Carriere M, Gosseries O, Laureys S, Chatelle C. Simplified evaluation of CONsciousness disorders (SECONDs) in individuals with severe brain injury: A validation study. Ann Phys Rehabil Med. 2021 Sep;64(5):101432. doi: 10.1016/j.rehab.2020.09.001. Epub 2021 Jul 28. PMID 32992025
- [Background] Bower J, Magee WL, Catroppa C, Baker FA. Content Validity and Inter-rater Reliability of the Music Interventions in Pediatric DoC Behavior Observation Record. J Music Ther. 2023 May 5;60(1):13-35. doi: 10.1093/jmt/thac013. PMID 36197798